CLINICAL TRIAL: NCT00138801
Title: Effect of Intravenous Ceftriaxone and Oral Doxycycline for Lyme Neuroborreliosis. A Randomized Double-blind Comparison
Brief Title: Effect of Intravenous Ceftriaxone and Oral Doxycycline for Lyme Neuroborreliosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: SSHF813204
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2005-03

CONDITIONS: Lyme Neuroborreliosis
Keywords: Neuroborreliosis
MeSH Terms: conditions — Lyme Neuroborreliosis | interventions — Ceftriaxone; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Doxycycline
  Interventions: Drug: Doxycycline
- 2 (Active Comparator): cephtriaxone
  Interventions: Drug: Ceftriaxone

INTERVENTIONS:
Drug: Ceftriaxone
  Arms: 2
Drug: Doxycycline
  Arms: 1

SUMMARY:
The aim of this study is to compare parenteral ceftriaxone and oral doxycycline in the treatment of neuroborreliosis in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Neurological symptoms and/or findings consistent with neuroborreliosis and at least one of the following fulfilled:

  * Intrathecal production of borrelia antibodies;
  * White cell count in cerebrospinal fluid (CSF) > 5/mm3;
  * Significant rise in borrelia antibodies in two serum samples collected from a patient with at least 3 weeks interval;
  * Verified acrodermatitis chronica atrophicans.

Exclusion Criteria:

* Allergy to the contents in the medication, or earlier type I reaction to penicillin.
* Treatment with cephalosporins, penicillin or tetracyclins during the last 14 days
* Pregnancy or breastfeeding
* Age < 18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-03; Primary Completion 2008-03 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Åse Mygland, MD, PhD, Study Chair — Sorlandet Sykehus HF
Locations (1):
- Sørlandet Sykehus HF, Kristiansand, Vest-Agder, Norway

REFERENCES:
- [Derived] Ljostad U, Skogvoll E, Eikeland R, Midgard R, Skarpaas T, Berg A, Mygland A. Oral doxycycline versus intravenous ceftriaxone for European Lyme neuroborreliosis: a multicentre, non-inferiority, double-blind, randomised trial. Lancet Neurol. 2008 Aug;7(8):690-5. doi: 10.1016/S1474-4422(08)70119-4. Epub 2008 Jun 21. PMID 18567539